CLINICAL TRIAL: NCT06311747
Title: The Immediate Effect of Including Oculo-motor Exercises in the Warm-up on Forehand and Backhand Stroke Performance in Tennis Players
Brief Title: The Effect of Oculomotor Exercises in the Warm-up on Forehand and Backhand Stroke Performance in Tennis Players
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Cim Cinar, Resident physician of Sports Medicine Department, Ege University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-1T/45
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Supportive Care
Keywords: Tennis; Oculomotor exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oculo-motor exercise (Experimental): Additional oculo-motor exercises will be administered to participants' warm-up before forehand and backhand stroke evaluation. As oculo-motor exercises, 3 different exercises will be applied: stepping exercise with eye movements and head rotation (The eyes are fixed on the thumb and the head rotates right and left and walks 10 steps forward and 10 steps back.), accommodation (First eyes fixed on the near target, then fixed on a target approximately 20-30 m away.) and pen tracking with 5 different movements (Horizontal, vertical, diagonal, circular, infinite eight).
  Interventions: Behavioral: Oculo-motor exercises

INTERVENTIONS:
Behavioral: Oculo-motor exercises — Oculo-motor exercises will be applied as an intervention. As oculo-motor exercises, 3 different exercises will be applied: stepping exercise with eye movements and head rotation (The eyes are fixed on the thumb and the head rotates right and left and walks 10 steps forward and 10 steps back.), accommodation (First eyes fixed on the near target, then fixed on a target approximately 20-30 m away.) and pen tracking with 5 different movements (Horizontal, vertical, diagonal, circular, infinite eight).

SUMMARY:
30 tennis players aged 12-18, will be included in the study. After their normal warm-up, the participants will make 30 forehand and 30 backhand strokes. Forehand and backhand stroke accuracy rate will be calculated. After a week, additional oculo-motor exercises will be included in the warm-up and the forehand and backhand stroke accuracy rate will be calculated again. The hypothesis that there will be an improvement in forehand and backhand stroke accuracy after oculo-motor exercises will be tested.

DETAILED DESCRIPTION:
30 tennis players aged 12-18, who practice tennis for at least 6 hours a week and have been playing regularly for at least 1 year will be included in the study. The positive effect of oculo-motor exercises to be included in the pre-tennis warm-up program on stroke performance will be investigated. As oculo-motor exercises, 3 different exercises will be applied: stepping exercise with eye movements and head rotation (The eyes are fixed on the thumb and the head rotates right and left and walks 10 steps forward and 10 steps back.), accommodation (First eyes fixed on the near target, then fixed on a target approximately 20-30 m away.) and pen tracking with 5 different movements (Horizontal, vertical, diagonal, circular, infinite eight). Participants will be given a backhand and forehand stroke evaluation consisting of a total of 60 strokes, 30 forehand and 30 backhand. In the first evaluation, the participants will be asked to do their regular warm-up program. The area between the baseline line, service line and singles side line on the tennis court will be marked and two target areas will be created, one on the right and one on the left. Players will be asked to take one stroke parallel and one stroke diagonally, and they will be expected to hit the marked target areas. One week later there will be a second evaluation. In the second evaluation, oculo-motor exercises will be included in the participants' warm-up programs and the stroke evaluation will be repeated. The data obtained will be evaluated whether oculo-motor exercises have a positive effect on the forehand and backhand stroke rate.

ELIGIBILITY:
Inclusion Criteria:

* Being 12-18 years old
* Playing tennis for at least 6 hours a week
* Having been playing tennis for at least 1 year
* No visual defect (myopia, hyperopia, astigmatism)

Exclusion Criteria:

* Being under 12 years old
* Being over 18 years old
* Playing tennis for less than 6 hours a week
* The duration of playing tennis is less than 1 year
* Having visual impairment (myopia, hyperopia, astigmatism)

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Forehand and backhand stroke accuracy | baseline and week 1
  30 forehand strokes and 30 backhand strokes will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Cengizhan OZGURBUZ, Study Director — Ege University Medical Faculty Hospital. Department of Sports Medicine; Cim CINAR, Principal Investigator — Ege University Medical Faculty Hospital. Department of Sports Medicine
Locations (1):
- Ege University Sports Medicine Clinic, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leith RJ, Zee DS: The Neurology of Eye Movements. Philadelphia, FA Davis, 1991, ed 2
- [Background] Gao Y, Chen L, Yang SN, Wang H, Yao J, Dai Q, Chang S. Contributions of Visuo-oculomotor Abilities to Interceptive Skills in Sports. Optom Vis Sci. 2015 Jun;92(6):679-89. doi: 10.1097/OPX.0000000000000599. PMID 25930979
- [Background] Pienaar, A.E. Motoriese Ontwikkeling, Groei, Motoriese Agterstande, die Assessering en Intervensie Daarvan: N Handleiding vir Nagraadse Studente in Kinderkinetika (Motor Development, Growth, Motor Delays, the Assessment and Intervention Thereof: A Guide for Post-Graduate Students); Xerox: Potchefstroom, South Africa, 2019; pp. 195?370.
- [Background] Marieb EN, Mallatt J. Human anatomy. California: Benjamin Cummings; 1992, p. 415?423.
- [Background] Williams AM, Ford PR. Expertise and expert performance in sport. Int Rev Sport Exerc Psychol 2008;1:4?18.
- [Background] Bouchard, D.; Tetreault, S. The motor development of sighted children and children with moderate low vision aged 8-13 J. Vis.Impair. Blind. 2000, 94, 564-573.
- [Background] Graybiel, A. (1955). Russian studies in vision in relation to physical activity and sports. Research Quarterly for Sports and Exercise, 26, 212-2.
- [Background] Garner AI. Scoring with sports vision. Optometric Management Magazine. 1985;21(8):24-32.
- [Background] Ripoll, H., & Fleurance, P. (1987). Dynamic Visual activity and eye movements: From physiology to cognition. Amsterdam: Elsevier. (p. 616-619).
- [Background] Rösblad, B.; Von Hofsten, C. Repetitive goal-directed arm movements in children with developmental coordination disorders: Role of visual information. Adapt. Phys. Activ. Q. 1994, 11, 190?202.
- [Background] Mann DL, Spratford W, Abernethy B. The head tracks and gaze predicts: how the world's best batters hit a ball. PLoS One. 2013;8(3):e58289. doi: 10.1371/journal.pone.0058289. Epub 2013 Mar 13. PMID 23516460
- [Background] Krüger, P.E.; Capher, J.; Smit, C.E. The role of visual skills and its impact on skill performance of cricket players. Afr. J. Phys. Health Educ. Recreat. Danc. 2009, 15, 605?623.
- [Background] Minoonejad H, Barati AH, Naderifar H, Heidari B, Kazemi AS, Lashay A. Effect of four weeks of ocular-motor exercises on dynamic visual acuity and stability limit of female basketball players. Gait Posture. 2019 Sep;73:286-290. doi: 10.1016/j.gaitpost.2019.06.022. Epub 2019 Jul 16. PMID 31398634
- [Background] Abernethy B, Wood JM. Do generalized visual training programmes for sport really work? An experimental investigation. J Sports Sci. 2001 Mar;19(3):203-22. doi: 10.1080/026404101750095376. PMID 11256825
- [Background] Amr H. A specific Visual Skills Training Programme Improves Fencing Performance Level, Visual Variables and Statics Balance,10th Annual Congress of the European College of Sport Since, Belgrade,316 ,2005.
- [Background] Bressan, E. S. (2003). Effects of visual skills training, vision coaching and sports vision dynamics on the performance of a sport skill. African Journal for Physical, Health Education, Recreation and Dance, 9(1), 20-31.
- [Background] Strainchamps P, Ostermann M, Mierau A, Hulsdunker T. Stroboscopic Eyewear Applied During Warm-Up Does Not Provide Additional Benefits to the Sport-Specific Reaction Speed in Highly Trained Table Tennis Athletes. Int J Sports Physiol Perform. 2023 Jun 15;18(10):1126-1131. doi: 10.1123/ijspp.2022-0426. Print 2023 Oct 1. PMID 37321564
- [Background] Cheatum, B.A.; Hammond, A.A. Physical Activities for Improving Children?s Learning and Behavior: A Guide to Sensory Motor Development; Human Kinetics: Champaign, IL, USA, 2000; pp. 185?263.
- [Background] Ferrauti A, Neumann G, Weber K, Keul J. Urine catecholamine concentrations and psychophysical stress in elite tennis under practice and tournament conditions. J Sports Med Phys Fitness. 2001 Jun;41(2):269-74. PMID 11447373
- [Background] Krzepota J, Zwierko T, Puchalska-Niedbal L, Markiewicz M, Florkiewicz B, Lubinski W. The Efficiency of a Visual Skills Training Program on Visual Search Performance. J Hum Kinet. 2015 Jul 10;46:231-40. doi: 10.1515/hukin-2015-0051. eCollection 2015 Jun 27. PMID 26240666
- [Background] Reimer, A.M.; Smits-Engelsman, B.C.M.; Siemonsma-Boom, M. Development of an instrument to measure manual dexterity in children with visual impairments aged 6?12. J. Vis. Impair. Blind. 2000, 94, 177?188.
- [Background] Huttermann S, Memmert D, Simons DJ. The size and shape of the attentional "spotlight" varies with differences in sports expertise. J Exp Psychol Appl. 2014 Jun;20(2):147-57. doi: 10.1037/xap0000012. Epub 2014 Apr 7. PMID 24708354
- [Background] Williams AM, Ward P, Knowles JM, Smeeton NJ. Anticipation skill in a real-world task: measurement, training, and transfer in tennis. J Exp Psychol Appl. 2002 Dec;8(4):259-70. doi: 10.1037//1076-898x.8.4.259. PMID 12570100
- [Background] Wilson, T.A.; Falkel, J. Sportsvision: Training for Better Performance; Human Kinetics: Champaign, IL, USA, 2004; p. 166.
- [Background] Sherman A. Overview of research information regarding vision and sports. J Am Optom Assoc. 1980 Jul;51(7):661-6. No abstract available. PMID 6995518
- [Background] Gonzalez-Gonzalez I, Rodriguez-Rosell D, Clavero-Martin D, Mora-Custodio R, Pareja-Blanco F, Garcia JMY, Gonzalez-Badillo JJ. Reliability and Accuracy of Ball Speed During Different Strokes in Young Tennis Players. Sports Med Int Open. 2018 Sep 25;2(5):E133-E141. doi: 10.1055/a-0662-5375. eCollection 2018 Sep. PMID 30539130
- [Background] Robinson DA: Control of eye movements, in Brooks VB (ed): Handbook of Physiology, Section 1, Tke Nervous System, Bethesda, American Physiological Society, 1981, pp 1275-1320
- [Background] Shim J, Carlton LG, Chow JW, Chae WS. The use of anticipatory visual cues by highly skilled tennis players. J Mot Behav. 2005 Mar;37(2):164-75. doi: 10.3200/JMBR.37.2.164-175. PMID 15730949
- [Background] Christenson GN, Winkelstein AM. Visual skills of athletes versus nonathletes: development of a sports vision testing battery. J Am Optom Assoc. 1988 Sep;59(9):666-75. PMID 3183281
- [Background] Erickson, G. B. (2007). Sports vision: Vision care for the enhancement of sports performance. St. Louis,MO: Butterworth-Heinemann.
- [Background] Buys JHC, Ferreira JT. The development of protocols and norms for sports vision evaluations. Afr Vision Eye Health. 2008;67(3):106?117. https://doi.org/10.4102/ aveh.v67i3.187
- [Background] S. Standring, Gray?s Anatomy: 7e Anatomical Basis of Clinical Practice, Churchill Livingstone, London, UK, 41st edition, 2016.
- [Background] Mendez-Villanueva A, Fernandez-Fernandez J, Bishop D, Fernandez-Garcia B, Terrados N. Activity patterns, blood lactate concentrations and ratings of perceived exertion during a professional singles tennis tournament. Br J Sports Med. 2007 May;41(5):296-300; discussion 300. doi: 10.1136/bjsm.2006.030536. Epub 2007 Jan 19. PMID 17237121